CLINICAL TRIAL: NCT05136417
Title: Safety and Feasibility of Intra-Cardiac Echocardiography in Guiding Left Atrial Appendage Occlusion With the Watchman Device: The ICE WATCHMAN Study
Brief Title: Study of Intra-Cardiac Echocardiography in Guiding Left Atrial Appendage Occlusion With the Watchman Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohamad Adnan Alkhouli, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-009613
Record Dates: First submitted 2021-11-25; First posted 2021-11-29 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Left Atrial Appendage Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- left atrial appendage (LAA) occlusion with the WATCHMAN FLX device using (ICE) (Experimental): 100 patients undergoing LAA closure with the WATCHMAN FLX utilizing an intra-procedural ICE probe under moderate sedation.
  Interventions: Device: intra-procedural intracardiac echocardiography (ICE) probe

INTERVENTIONS:
Device: intra-procedural intracardiac echocardiography (ICE) probe — placing the WATCHMAN FLX device using the intra-procedural intracardiac echocardiography (ICE) probe.

SUMMARY:
The purpose of this research is to to assess the feasibility and safety of left atrial appendage (LAA) occlusion with the WATCHMAN FLX™ device using a standardized intra-procedural intracardiac echocardiography (ICE) protocol under moderate sedation for procedural guidance.

ELIGIBILITY:
Inclusion Criteria:

* The patients is eligible to undergo WATCHMAN device implant procedure.
* The patient is eligible for short term anticoagulation therapy.
* Ability to tolerate the procedure without the need for general anesthesia as assessed by the treating physician(s).
* Ability to give informed consent for the procedure.
* The patient is able and willing to undergo the procedure under moderate sedation.
* The patient is able and willing to return for required 45-day transesophageal echocardiogram (TEE).

Exclusion Criteria:

* Patient has contraindication for short term anticoagulation.
* The patient has history of a hypercoagulable state per medical record documentation.
* Pregnancy or planning to get pregnant during the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Adnan Alkhouli, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Pacific Heart Institute, Santa Monica, California
  - Mayo Clinic in Rochester, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE): 100 patients undergoing left atrial appendage (LAA) closure with the WATCHMAN FLX utilizing an intra-procedural ICE probe under moderate sedation.
  intra-procedural intracardiac echocardiography (ICE) probe: placing the WATCHMAN FLX device using the intra-procedural intracardiac echocardiography (ICE) probe.
Period: Overall Study
Arm/Group | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE)
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE)
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Successful Implantation of WATCHMAN FLX Device
Description: Number of participants with a successfully implanted WATCHMAN FLX device. Implant success is defined as confirmation of the device-specified release PASS (Position, Anchor, Size, Seal) criteria, successful device release, and adequate seal (defined as a residual leak <5 mm) as assessed by a core lab interpretation of the transesophageal echocardiogram (TEE) 45 days post-implant.
Time Frame: 45 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE)
Number analyzed (Participants) | 100
Participants | 96

2. Primary Outcome: Major Complications
Description: Number of participants who experience major complications defined as major bleeding (intracranial bleeding, or bleeding requiring blood transfusion), pericardial effusion requiring pericardiocentesis or surgery, device embolization, procedural-related stroke, or procedural related death).
Time Frame: up to 7 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE)
Number analyzed (Participants) | 100
Participants | 3

3. Secondary Outcome: Procedure Conversion to General Anesthesia
Description: Number of participants who required conversion from moderate sedation to general anesthesia for implant procedure.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE)
Number analyzed (Participants) | 100
Participants | 0

4. Secondary Outcome: Iatrogenic Atrial Septal Defect
Description: Number of participants with an iatrogenic atrial septal defect.
Time Frame: 45 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE)
Number analyzed (Participants) | 100
Participants | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each participant from enrollment to 45 days post procedure, for a total of approximately 60 days.
Arm/Group | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE)
All-Cause Mortality (participants affected / at risk) | 1/100
Serious Adverse Events (participants affected / at risk) | 3/100
Other Adverse Events (participants affected / at risk) | 10/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE) (N=100)
Gastrointestinal bleeding requiring transfusion (Gastrointestinal disorders) | 2 (2)
Procedural-related stroke (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Left Atrial Appendage (LAA) Occlusion With the WATCHMAN FLX Device Using (ICE) (N=100)
Access site hematoma (General disorders) | 5 (5)
Postoperative bleeding (General disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT05136417/Prot_000.pdf